CLINICAL TRIAL: NCT03201640
Title: Virtual Reality for Educating and Reducing Preoperative Anxiety in Children - A Randomised Control Trial
Brief Title: VR for Preoperative Anxiety in Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Hospital for Sick Children (Other)
Responsible Party: Principal Investigator, Clyde Matava, Staff Anesthesiologist, The Hospital for Sick Children
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 1000056779
Record Dates: First submitted 2017-06-26; First posted 2017-06-28 (Actual); Last update posted 2021-12-17 (Actual); Status verified 2021-12

CONDITIONS: Anxiety
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- slideshow (Other): Participant receives traditional slideshow presentation for preoperative preparation
  Interventions: Behavioral: slideshow
- virtual (Other): Participant receives virtual reality presentation for preoperative preparation
  Interventions: Behavioral: virtual

INTERVENTIONS:
Behavioral: slideshow — Participants will be shown a slideshow showing a child being prepared for surgery
  Arms: slideshow
Behavioral: virtual — Participants will be shown an immersive virtual reality preparation for surgery
  Arms: virtual

SUMMARY:
All of the tools currently available for preoperative preparation of children either use a third person approach (i.e., use media whereby they watch a video or look at pictures of another child receiving an anesthetic), provide tours at some time previous to the operation date, or are shown the equipment that they will encounter during their anesthetic. No preoperative programme currently allows the child to experience the entire chain of events from leaving the preoperative preparation area (and their parents), walking to the operating area, being initially prepared for and receiving anesthesia and recovering from anesthesia, in real time and from a first person perspective. As such the investigators are carrying out this study to assess whether virtual reality preoperative preparation is effective in reducing anxiety at induction of anesthesia.

DETAILED DESCRIPTION:
The investigators' goal in this study is to investigate the effects of virtual reality preoperative preparation on anxiety in children at induction of anesthesia. The hypothesis is that utilisation of this novel 1st person immersive preparatory method will lead to an enhanced understanding of what will happen to the child (in addition to what the environment looks and sounds like) when they have their anesthetic. The investigators believe this enhanced understanding and preparation will lead to the reduction in anxiety levels before and during the induction of anesthesia, and will also lead to a reduction in postoperative negative behaviour disorders.

ELIGIBILITY:
Inclusion Criteria:

1. Patients aged between 6 -18
2. ASA physical status 1-3
3. Admitted for elective surgery (day case and inpatient cases)
4. Cognitively normal

Exclusion Criteria:

1. ASA physical status 4-5
2. Non-English speaking
3. Significant visual and auditory disorders not allowing them to use the technology
4. Epilepsy
5. Mobility problems that would make using the technology difficult or harmful to them (i.e., reduced movement of neck)
6. Cognitive impairment
7. Postoperative PICU care anticipated

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 39 (Actual)
Dates: Start 2017-09-18 (Actual); Primary Completion 2019-04-30 (Actual); Study Completion 2019-04-30 (Actual)

PRIMARY OUTCOMES:
Anxiety in children | Day of surgery, immediately following consent
  measured using the modified Yale Preoperative Anxiety Scale (mYPAS)
Change in child anxiety | Day of surgery, immediately preceding surgery
  measured using the modified Yale Preoperative Anxiety Scale (mYPAS)

SECONDARY OUTCOMES:
Induction compliance | Day of surgery, immediately preceding surgery
  measured using the Induction Compliance Checklist
Anesthetic requirements | Day of surgery, intra-operatively
  measurement includes recording dose of anesthetic(s) used
Post-hospitalization negative behaviours | Two to three days after surgery
  measured using the Posthospitalization Behaviour Questionnaire (PHBQ)

CONTACTS AND LOCATIONS:
Overall Officials: Clyde Matava, Principal Investigator — The Hospital for Sick Children
Locations (1):
- The Hospital for Sick Children, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No